CLINICAL TRIAL: NCT03915795
Title: Application of Statins in Long-term Treatments of Kawasaki Disease Complicated With Severe Coronary Artery Abnormalities in Children
Brief Title: Statins Study in Kawasaki Disease Children With Coronary Artery Abnormalities
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: Statins study in KD
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Kawasaki Disease; Coronary Artery Abnormalities
Keywords: Kawasaki Disease; coronary artery abnormalities; statins
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the effects of statins on chronic inflammation, coronary artery abnormalities and clinical cardiac events in long-term KD children complicated with severe coronary artery abnormalities, and the feasibility and safety of statins in treatment of KD children.

DETAILED DESCRIPTION:
Kawasaki disease (KD) is an acute self-limited vasculitis and occurs almost exclusively in childhood. It predominantly affects medium-sized arteries, most commonly the coronary arteries. Although the use of intravenous immunoglobulin (IVIG) has obviously decreased the incidence of coronary arteries (CA) abnormalities, still a part of KD children occur CA abnormalities, even medium, large or giant aneurysms. The coronary aneurysms can develop to thrombus and arterial stenosis, which may cause severe cardiac events, for example, myocardial infarction. It is the main cause of disability and death in KD children. Now KD has been the leading cause of acquired heart disease in children.

Some studies found that ongoing vascular chronic inflammation and oxidative stress persisted in the long-term KD vasculopathy. Endothelial dysfunction, increased stiffness, and intima-media thickening have been noted in both affected coronary arteries and systemic arteries. Statins (hydroxymethylglutaryl coenzyme-A reductase inhibitors) not only are a kind of drug lowering low-density lipoprotein cholesterol, but also have been reported to have potentially beneficial pleiotropic effects on inflammation, endothelial function, oxidative stress, platelet aggregation, coagulation, and fibrinolysis. They have been the cornerstone of therapy for the primary and secondary prevention of atherosclerotic cardiovascular events in adults. In recently years, statins have been considered to be used in KD children with coronary aneurysms. Several short-term small studies in such patients treated with statins have shown reductions in high-sensitivity CRP, improved endothelial function and statins' safety in children. The American Heart Association (AHA) scientific statement on KD published in 2017 suggests that empirical treatment with low-dose statin may be considered for KD patients with past or current aneurysms, regardless of age or sex.

However, the current clinical data about the use of statins in KD children is still very rare. The published researches mainly focused on the endothelial function of peripheral arteries but the effects of statins on CAs and cardiac events have not been included. Therefore, more studies are needed to conform statins' feasibility and safety in children and its clinical application value.

In this study, we will recruit KD children complicated with severe CA abnormalities. These children will be given statins for one year besides other routine treatments. The coronary assessments, clinical and laboratory indexes will be followed up to study the effects of statins on long-term chronic inflammation, CA abnormalities and clinical cardiac events. At the same time, the clinical and laboratory indexes correlated to the side-effects will be monitored regularly to investigate the feasibility and safety of statins in KD children.

ELIGIBILITY:
Inclusion Criteria:

* >3 months after the onset of KD currently complicated with severe coronary artery abnormalities (medium coronary aneurysms or more severe) The follow-up can be achievable All included children's guardian are required to sign the informed consent form

Exclusion Criteria:

* The KD children currently complicated with mild coronary artery abnormalities (small aneurysms or only dilation) The children's age <2 ys The children's guardian don't agree to sign the informed consent

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The KD children admitted to the Cardiology ward in Children's Hospital of Fudan University, Shanghai, China
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change of coronary artery abnormalities measured by echocardiography | At baseline and one year after taking statin
  Internal lumen diameters(mm) and Z score of coronary artery abnormalities measured by echocardiography

SECONDARY OUTCOMES:
Change of LDL-C | At baseline and one year after taking statin
  Decrease in LDL-C(mmol/L)
Change of high-sensitivity C reactive protein (hsCRP) | At baseline and one year after taking statin
  Decrease in hsCRP (mg/L) as a chronic inflammation marker
Assessment of myocardial ischemia | At baseline and one year after taking statin
  New onset or improved manifestation of myocardial ischemia, assessed by EKG/stress EKG, radionuclide myocardial imaging and/or magnetic resonance imaging
Incidence of new-onset cardiovascular events | One year after taking statin
  Incidence of new-onset cardiovascular events including chest tightness, chest pain, angina, myocardial infarction and so on
Incidence of side-effects of statin in KD children | At baseline, 3, 6, 9 months and one year after taking statins
  Incidences of side-effects including abnormal laboratory indexes (elevated muscle enzyme and liver enzyme), adverse clinical events and growth impacts (weight, height and BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Fang Liu, MD, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No